CLINICAL TRIAL: NCT01724775
Title: A Prospective, Non-randomized, Double-blind, Single-center Study to Evaluate Efficacy and Safety of Complete Mesocolic Excision for Colon Cancer.
Brief Title: Efficacy and Safety Study of Complete Mesocolic Excision for Colon Cancer
Acronym: ESCME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shan Wang (Other)
Responsible Party: Sponsor-Investigator, Shan Wang, Department of Gastrointestinal Surgery, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: PKPH-CME; Z121100005312015 (Other Grant/Funding Number: Science and Technology Project of Bejing, China); TG-2015-002 (Other Grant/Funding Number: Capital health development research project); 20130001120064 (Other Grant/Funding Number: Doctoral Program of Higher Education)
Record Dates: First submitted 2012-11-04; First posted 2012-11-12 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Colon Cancer; Surgery
Keywords: complete mesocolic excision; colon cancer; efficacy; safety
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CME surgery for colon cancer
- non-CME surgery for colon cancer

SUMMARY:
In 2009, Prof. Hohenberger proposed complete mesocolic excision (CME) as standardized, in which the same principle of TME in rectal cancer has been applied to the colon. More and more surgeons pay attention to the rationality of this surgical approach. However, the clinical application researches are still few, in particular the prospective controlled study is still none. This clinical trial will compare the CME group and non-CME group to evaluate the outcome and safety of CME for apply in clinic.

DETAILED DESCRIPTION:
Materials and Methods:

All the patients with colon cancer will undergo elective radical operation. The observations were recorded during the operation and on the postoperative specimens. Intra-operative photographs were taken at various stages, as were photographs of the postoperative specimen. According to the CME operation keypoints, all the photographs will accept third-party assessment of the expert group, while the third-party expert group will not participate in the management of patients. Both of The evaluators and research doctors are double-blind state. The postoperative patients will divided into two groups according to the results of the assessment. The clinical and pathological data of the patients as well as follow-up information will be recorded and collected.

1. Outcome of CME By comparison to clinicopathologic variables, and precise tissues morphometry of two groups, the prognosis, lymph nodes harvest and removal of the mesocolic area were investigated. Outcomes of interest also include disease-free survival, local recurrence-free survival, recurrence rate. In addition, we analyzed the correlation between mesocolic area and height, weight, body surface area and body mass index.
2. Safety of CME CME group and non-CME group were compared the differences of security, included operation time, blood loss, postoperation complications, flatus restoring time, defecation restoring time, drainage removal time, Diet restoring time, drainage volume in three days after surgery, hospital deaths, the exhaust time, hospitalization time and hospitalization costs. In addition, the feasibility of CME techniques as the surgical approach of choice for elderly patients was also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of colon cancer;
* Clinical stage Ⅰ ~ Ⅲ;
* Undergoing colorectal surgery for the first time;
* Accept laparotomy;
* Accept radical resection;
* More than 18 years.

Exclusion Criteria:

* Emergency surgery;
* Preoperative neoadjuvant chemoradiotherapy history;
* Combined with other malignant diseases;
* Pathological stage Ⅳ patients with colon cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of colon caner in China
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2012-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Prognosis assessment of postoperative patients | yearly, up to 5 years
  The assessment of 5-year and 3-year overall survival, disease-free survival, local recurrence rate, local recurrence-free survival for postoperative patients respectively.

SECONDARY OUTCOMES:
Safety assessment of the patients in perioperation period | Daily, up to one month
  Includes: postoperative complications, hospital mortality, operative time, blood loss, exhaust time, defecation time, drainage and unplug time, resumed eating time, drainage volume during postoperation three days and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Yingjiang Ye, M.D. & Ph.D., Study Director — Peking University People's Hospital
Locations (1):
- Department of Gastroenterology Surgery, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang C, Gao Z, Shen Z, Jiang K, Zhou J, Wang S, Ye Y. Five-Year Prognosis of Complete Mesocolic Excision in Patients with Colon Cancer: A Prospective, Nonrandomized, Double-Blind Controlled Trial. J Am Coll Surg. 2022 Oct 1;235(4):666-676. doi: 10.1097/XCS.0000000000000282. Epub 2022 Sep 15. PMID 36106868
- [Derived] Gao Z, Wang C, Cui Y, Shen Z, Jiang K, Shen D, Wang Y, Zhan S, Guo P, Yang X, Liu F, Shen K, Liang B, Yin M, Xie Q, Wang Y, Wang S, Ye Y. Efficacy and Safety of Complete Mesocolic Excision in Patients With Colon Cancer: Three-year Results From a Prospective, Nonrandomized, Double-blind, Controlled Trial. Ann Surg. 2020 Mar;271(3):519-526. doi: 10.1097/SLA.0000000000003012. PMID 30148752